CLINICAL TRIAL: NCT07282158
Title: Adaptation of Helping Ovarian Cancer Patients Cope (HOPE) for Clinician Burnout (HOPE-C)
Brief Title: Adapted Helping Ovarian Cancer Patients Cope Intervention to Address Burnout for Gynecologic Oncology Clinicians
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: Andy Hill CARE Fund (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: RG1125922; NCI-2025-07869 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); FHIRB0021069 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2025-12-01; First posted 2025-12-15 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2025-12

CONDITIONS: Ovarian Carcinoma; Psychiatric Disorder
MeSH Terms: conditions — Ovarian Neoplasms; Mental Disorders | interventions — Behavior Therapy; Memory and Learning Tests; Interviews as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HOPE-C intervention (Experimental): OBJECTIVE 1 DEVELOPMENT OF INTERVENTION: Clinicians review HOPE-C intervention materials and complete an interview and questionnaire on study. Feedback from Objective 1 will be incorporated into the HOPE-C intervention delivered in Objective 2.
  OBJECTIVE 2 PILOT TRIAL: Clinicians attend HOPE-C sessions (changing their narrative, managing life's uncertainty and finding meaning) once weekly for 4 weeks, with each session lasting approximately 30-45 minutes. Clinicians complete a questionnaire before and after completing all HOPE-C sessions.
  OBJECTIVE 3: Clinicians may undergo an interview after completing HOPE-C sessions.
  Interventions: Behavioral: Behavioral Intervention; Other: Interview; Other: Survey Administration

INTERVENTIONS:
Behavioral: Behavioral Intervention — Complete HOPE-C sessions
  Other Names: Behavior Conditioning Therapy; Behavior Modification; Behavior or Life Style Modifications; Behavior Therapy; Behavioral Interventions; Behavioral Modification; Behavioral Therapy; Behavioral Treatment; Behavioral Treatments; Behavioural
Other: Interview — Complete interview
Other: Survey Administration — Ancillary studies

SUMMARY:
This clinical trial tests an adapted version of the Helping Ovarian Cancer Patients Cope (HOPE) intervention to address burnout among gynecologic oncology clinicians. Stress and burnout among gynecologic oncology clinicians can have far-reaching impacts not only on physicians at the individual level (e.g., distress, mental illness) but also at the professional (e.g., worse patient outcomes, increased errors) and societal levels (fewer physicians in this specialty, more system strain). The original Helping Ovarian Cancer Patients Cope (HOPE) is a workshop to promote hope among patients with ovarian cancer through creating positive narratives using the hope theory and social-cognitive theory. The adapted intervention for clinicals (HOPE-C) will use the same concepts but tailored to clinician experiences by fostering peer support and retelling their challenging stories and may address burnout for gynecologic oncology clinicians.

DETAILED DESCRIPTION:
OUTLINE:

OBJECTIVE 1 DEVELOPMENT OF INTERVENTION: Clinicians review HOPE-C intervention materials and complete an interview and questionnaire on study.

OBJECTIVE 2 PILOT TRIAL: Clinicians attend HOPE-C sessions (changing their narrative, managing life's uncertainty and finding meaning) once weekly for 4 weeks, with each session lasting approximately 30-45 minutes. Clinicians complete a questionnaire before and after completing all HOPE-C sessions.

OBJECTIVE 3: Clinicians may undergo an interview after completing HOPE-C sessions.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years of age or older
* English speaking
* Able to provide informed consent
* Working with patients with ovarian cancer (gynecologic oncologists, medical oncologists, nurses, social workers, and advance practice providers [APPs])

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective 1: Clinician feedback for Helping Ovarian Cancer Patients Cope-Clinician Burnout (HOPE-C) | Day 1
  Will assess clinician's feedback around the content, delivery structure, and materials for the adapted HOPE-C intervention. Qualitative Description will be used to analyze the data.
Objective 2: Feasibility (Accrual rate) | At time of enrollment
  Feasibility cutoff includes ≥ 50% of eligible clinicians enrolling in the study.
Objective 2: Feasibility (Rate of intervention completion) | At 4 weeks
  Feasibility cutoff includes ≥ 50% of enrolled clinicians completing all sessions.
Objective 2: Feasibility (Rate of survey completion) | At baseline and 2-week post-intervention
  Feasibility cutoff includes ≥ 50% of enrolled clinicians completing all surveys.
Objective 2: Acceptability of HOPE-C | At 2-week post-intervention
  Assessed by the Theoretical Framework of Acceptability (TFA) questionnaire, which is an 8-item questionnaire assessing acceptability of healthcare interventions across seven constructions: Affective Attitude, Burden, Ethicality, Intervention Coherence, Opportunity Costs, Perceived Effectiveness and Self-efficacy. Items are rated on a 5-point Likert scale (e.g., 1 = strongly dislike, 5 = strongly like) and a mean is computed across all seven constructs (n=7 items) and a single outcome is examined for the general item. Total mean score ranges from 1 to 5, with higher scores indicating greater acceptability of the intervention.
Objective 2: Satisfaction of HOPE-C | At 2-week post-intervention
  Will be assessed by using three items assessing overall satisfaction. A cutoff score of ≥ 7 (out of 10) will be used for each satisfaction item.
Objective 3: Optimization of the intervention | At 2-week post-intervention
  Feedback will be gathered from clinicians who participated in the intervention to assess their feedback on how to optimize the intervention in clinical settings.
Objective 3: Delivery of the intervention | At 2-week post-intervention
  Feedback will be gathered from clinicians who participated in the intervention to assess their feedback on the delivery of the intervention in clinical settings.

CONTACTS AND LOCATIONS:
Overall Officials: Megan J. Shen, PhD, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No